CLINICAL TRIAL: NCT02922725
Title: A Randomized, Double-blind, Placebo-controlled Trial of 5-hydroxytryptophan and Creatine for SSRI or SNRI Augmentation in Treatment Resistant Depression Associated With Hypobaric Hypoxia in Females
Brief Title: Placebo-controlled Trial of 5-hydroxytryptophan and Creatine for SSRI or SNRI Augmentation in Treatment Resistant Depression in Females
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: Brent Michael Kious, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Brent Michael Kious, MD, PhD, Instructor, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 94176
Record Dates: First submitted 2016-09-28; First posted 2016-10-04 (Estimated); Results first posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — 5-Hydroxytryptophan; Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Depressed patients receiving study drug (Active Comparator): Participants diagnosed with MDD
  Interventions: Drug: 5-hydroxytryptophan and Creatine
- Depressed patients receiving placebo (Placebo Comparator): Participants diagnosed with MDD
  Interventions: Other: Placebo control
- Healthy Control (No Intervention)

INTERVENTIONS:
Drug: 5-hydroxytryptophan and Creatine
  Arms: Depressed patients receiving study drug
Other: Placebo control
  Arms: Depressed patients receiving placebo

SUMMARY:
The investigators propose to determine if 8 weeks of dietary augmentation with oral 5g creatine monohydrate daily and 100 mg of 5-hydroxytryptophan (5-HTP) twice daily reduces hypoxia-related depressive symptoms measured by the 17-item Hamilton Depression Rating Scale (HAM-D) in women with SSRI- or SNRI-resistant depression, combined with the examination of changes in functional connectivity based on resting-state fMRI and changes in brain metabolism inferred from phosphorus-31 magnetic resonance spectroscopy.

DETAILED DESCRIPTION:
Serotonin and creatine are processed separately in the brain, and deficits in these brain biochemicals lead to distinct clinical problems. Therefore, investigators believe that treatment with a combination therapy, which could correct both deficits, would have a synergistic effect in the treatment of hypoxia-related depression and possibly other forms of treatment-resistant depression. Thus, investigators propose to investigate antidepressant efficacy of dietary 5-hydroxytryptophan (5-HTP) and creatine, as a means to restore the brain neurotransmitter and metabolic imbalances linked to chronic hypoxia caused by high altitude residence.

ELIGIBILITY:
Inclusion Criteria:

* Female gender, ages 25-40 years inclusive
* Current diagnosis of Major Depressive Disorder identified by the SCID-I
* Current HAM-D17 score of > 16
* Adequate adherence to any FDA approved SSRI or SNRI for at least 8 weeks
* Right-handed

Healthy Controls Inclusion criteria:

* Female gender, ages 25-40 inclusive
* No current or past DSM-5 diagnosis, as determined by clinical and structured interviews

Exclusion Criteria:

* Any non-MDD and non-anxiety psychiatric diagnosis, as identified by the SCID-I
* History of or current diagnosis of renal disease, such as chronic renal failure, acute renal failure or end stage renal disease
* Diabetes type I or II
* Current colitis or diverticulitis
* History of or current pulmonary disease
* History of cardiac disease or QTc > 500ms
* History of fibromyalgia, lupus, eosinophilia-myalgia syndrome, dermatomyositis, polymyositis, rheumatoid arthritis, psoriatic arthritis, mixed connective tissue disease, ankylosing spondylitis, or other related rheumatological condition
* History of or current seizure disorder
* Current serious suicide risk identified by the Columbia Severity Suicide Rating Scale
* Current treatment with an antipsychotic, mood stabilizer, or non-SSRI antidepressant
* Positive pregnancy test, pregnancy, failure to use adequate birth control method
* Previous diagnosis of serotonin syndrome or evidence of serotonin syndrome
* Use of any excluded drugs or medications including serotonergic drugs or medications (Table 2)
* Pre-existing eosinophilia (absolute eosinophil count > 500/uL)
* Contraindications to MRI: ferromagnetic implants, implanted devices, claustrophobia

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Depressed Patients Receiving Study Drug: Participants diagnosed with MDD
  5-hydroxytryptophan 100mg PO BID and Creatine monohydrate 5g PO Qday
- Depressed Patients Receiving Placebo: Participants diagnosed with MDD
  Placebo control (fructose 100mg PO BID and fructose 5g PO Qday)
- No Intervention: Healthy Controls: Healthy controls (no history of depression) recruited for neuroimaging comparison group
Period: Overall Study
Arm/Group | Depressed Patients Receiving Study Drug | Depressed Patients Receiving Placebo | No Intervention: Healthy Controls
Started | 12 | 12 | 8
Completed | 11 | 12 | 8
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Depressed Patients Receiving Study Drug: Participants diagnosed with MDD
  5-hydroxytryptophan and Creatine
- Depressed Patients Receiving Placebo: Participants diagnosed with MDD
  Placebo control
- Healthy Controls: Participants with no history of MDD
  No intervention
- Total: Total of all reporting groups
Arm/Group | Depressed Patients Receiving Study Drug | Depressed Patients Receiving Placebo | Healthy Controls | Total
Number analyzed (Participants) | 11 | 12 | 8 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 8 | 31
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 8 | 31
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 11 | 12 | 8 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 12 | 8 | 31
17-Item Hamilton Depression Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The total Hamilton Depression (HAM-D) Rating Scale provides and indication of depression
  In general, the higher the total score the more severe the depression.
  HAM-D score level of depression:
  10 - 13 mild; 14-17 mild to moderate; >17 moderate to severe.
  Range: 0 to 54 Population: Healthy controls were not asked to complete the depression measure (HAMD) because they did not have depression.
  units on a scale
    number analyzed (Participants) | 11 | 12 | 0 | 23
    (all) | 20.5 (3.4) | 20.1 (2.9) |  | 20.3 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hamilton Depression Rating Scale
Description: The total Hamilton Depression (HAM-D) Rating Scale provides and indication of depression In general, the higher the total score the more severe the depression.
  HAM-D score level of depression:
  10 - 13 mild; 14-17 mild to moderate; >17 moderate to severe. Range: 0 to 54
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Depressed Patients Receiving Study Drug | Depressed Patients Receiving Placebo
Number analyzed (Participants) | 11 | 12
units on a scale | 6.8 (5.5) | 7.3 (5.4)

ADVERSE EVENTS:
Time Frame: 8 weeks of study intervention with 4 weeks of post-treatment follow-up
Groups:
- Health Controls: Participants with no history of MDD
  No intervention
Arm/Group | Depressed Patients Receiving Study Drug | Depressed Patients Receiving Placebo | Health Controls
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/8

LIMITATIONS AND CAVEATS:
Difficulties with recruitment suggest that the study may have been underpowered to detect an effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/25/NCT02922725/Prot_SAP_000.pdf